CLINICAL TRIAL: NCT01897779
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single- and Multiple Ascending-dose Study of the Safety, Tolerability, and Pharmacokinetics of Intravenous RPX2014 and RPX7009 Alone and in Combination in Healthy Adult Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics of Intravenous RPX2014 and RPX7009 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rempex Pharmaceuticals (a wholly owned subsidiary of The Medicines Company) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rempex 501
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Volunteers; Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — RPX7009; beta-Lactamase Inhibitors; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Single and multiple dose of RPX7009 (Experimental): Single and multiple dose of RPX7009
  Interventions: Drug: RPX7009
- Single and multiple dose of RPX2014 (Experimental): Single and multiple dose of RPX2014
  Interventions: Drug: RPX2014
- Normal Saline (Placebo Comparator): Single and multiple dose of normal saline
  Interventions: Drug: Placebo
- Combination RPX7009 and RPX2014 (Experimental): Single and Multiple dose of Combination RPX7009 and RPX2014
  Interventions: Drug: Combination RPX7009 and RPX2014

INTERVENTIONS:
Drug: RPX7009 — Two (2) groups of 15 subjects (12 active and 3 placebo) are planned for evaluation in cohort 1. Cohorts 2-5, 14 subjects (11 active and 3 placebo) are planned for evaluation in each cohort. 14 subjects (12 active and 2 placebo) are planned for evaluation in cohort 6.
  Other Names: (beta-lactamase inhibitor)
  Arms: Single and multiple dose of RPX7009
Drug: RPX2014 — Two (2) groups of 15 subjects (12 active and 3 placebo) are planned for evaluation for cohort 1. Cohorts 2-5, 14 subjects (11 active and 3 placebo) are planned for evaluation in each cohort. 14 subjects (12 active and 2 placebo) are planned for evaluation in cohort 6.
  Arms: Single and multiple dose of RPX2014
Drug: Placebo — Two (2) groups of 15 subjects (12 active and 3 placebo) are planned for evaluation for cohort 1. Cohorts 2-5, 14 subjects (11 active and 3 placebo) are planned for evaluation in each cohort. 14 subjects (12 active and 2 placebo) are planned for evaluation in cohort 6.
  Other Names: Normal saline
  Arms: Normal Saline
Drug: Combination RPX7009 and RPX2014 — Two (2) groups of 15 subjects (12 active and 3 placebo) are planned for evaluation in cohort 1. Cohorts 2-5, 14 subjects (11 active and 3 placebo) are planned for evaluation in each cohort. 14 subjects (12 active and 2 placebo) are planned for evaluation in cohort 6.
  Arms: Combination RPX7009 and RPX2014

SUMMARY:
RPX7009 (beta-lactamase inhibitor) is being studied in combination with a carbapenem (RPX2014) to treat bacterial infections, including those due to multi-drug resistant bacteria.

DETAILED DESCRIPTION:
The worldwide spread of resistance to antibiotics among Gram-negative bacteria, particularly members of the ESKAPE group of pathogens, has resulted in a crisis in the treatment of hospital acquired infections. In particular, the recent dissemination of a serine carbapenemase (e.g., KPC) in Enterobacteriaceae in US hospitals now poses a considerable threat to the carbapenems and other members of the beta-lactam class of antimicrobial agents.

Rempex is developing a fixed combination antibiotic of a carbapenem (RPX2014) plus a new beta-lactamase inhibitor (RPX7009) which has activity against serine beta-lactamases, including KPC. This Phase 1 study will assess the safety, tolerability and pharmacokinetics of intravenous RPX2014 and RPX7009, administered alone and in combination, in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and females, 18 to 55 years of age (inclusive) at the time of screening.
2. Body mass index (BMI) ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive).
3. Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical histories, ECGs, physical examination) as deemed by the PI.
4. Non-tobacco/nicotine-containing product users for a minimum of Dose Study 6 months prior to Day 1.
5. Voluntarily consent to participate in the study.
6. Sexually abstinent or agree to use two approved methods of contraception.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
2. Positive urine drug/alcohol testing at screening or check-in (Day -1).
3. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
4. History or presence of alcoholism or drug abuse within the 2 years prior to Day 1.
5. Use of any over-the-counter (OTC) medication, including herbal products and vitamins, within the 7 days prior to Day 1. Up to 2 grams per day of acetaminophen is allowed for acute events at the discretion of the PI.
6. Blood donation or significant blood loss (i.e., > 500 mL) within 56 days prior to Day 1.
7. Plasma donation within 7 days prior to Day 1.
8. Participation in another investigational clinical trial within 30 days prior to Day 1.
9. Subjects who have any abnormalities on laboratory values at screening or check-in (Day -1).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety from baseline through the end of the study | Study Day 1 to Day 14
  Number of patients with adverse events; assessed by patient reporting, collection of vital signs, ECGs and absolute values and changes over time of hematology, chemistry and urinalysis.

SECONDARY OUTCOMES:
Composite of PK parameters RPX7009, RPX2014, combination of RPX7009 and RPX2014 & placebo following single and multiple dose administration. | Study Day1 to Day 14
  Plasma AUC0-t, AUC0-inf, Cmax, and Tmax.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Loutit, Study Director — Sponsor GmbH
Locations (1):
- CMAX, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Rubino CM, Bhavnani SM, Loutit JS, Morgan EE, White D, Dudley MN, Griffith DC. Phase 1 Study of the Safety, Tolerability, and Pharmacokinetics of Vaborbactam and Meropenem Alone and in Combination following Single and Multiple Doses in Healthy Adult Subjects. Antimicrob Agents Chemother. 2018 Mar 27;62(4):e02228-17. doi: 10.1128/AAC.02228-17. Print 2018 Apr. PMID 29437614